CLINICAL TRIAL: NCT05331508
Title: Testing the Integration of Gender-based Violence First-line Response in Family Planning and Antenatal Care Services in Nigeria
Brief Title: Testing Gender-based Violence Response in Family Planning and Antenatal Care Services in Nigeria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jhpiego (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCGL-IRB17494
Record Dates: First submitted 2022-02-28; First posted 2022-04-15 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Gender-based Violence; Reproductive Coercion; Intimate Partner Violence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Prior to commencement of the study, providers responsible for FP and ANC service provision will participate in a 3-day competency-based skills-building training activity on Caring for women subjected to violence: A WHO curriculum for training health-care providers and the ARCHES intervention. Following the training, providers will (1) introduce routine client screening for GBV, including intimate partner violence, sexual violence, and reproductive coercion using a standardized screening form, in FP and ANC services,(2) for individuals disclosing GBV, provide first-line response-empathetic counseling, including listening, inquiring about experiences sensitively, and validating experiences, helping clients develop safety plans, and providing support; (3) regardless of disclosure of GBV, provide counseling and information, education and communication (IEC) materials on IPV, including reproductive coercion, and FP options, to both FP and ANC clients.
  Interventions: Behavioral: gender-based violence screening, first-line support (LIVES) and reproductive coercion empowerment counseling (ARCHES)
- Control group (No Intervention): FP clients and ANC clients will receive standard care. For FP services, this includes standard contraceptive care provided by personnel who have completed training on contraceptive service delivery by the Nigerian Federal Ministry of Health and partners. For ANC services, the standard is a minimum of 8 visits with health personnel trained on ANC care during pregnancy. This includes identification of women and girls at increased risk of developing complications during labor and childbirth; prevention, detection, and management of pregnancy-related and concurrent conditions; health education and promotion; promotion of the use of skilled attendance at birth and healthy behaviors such as breastfeeding, early postnatal care, and planning for optimal pregnancy spacing, routine examinations, detection of complications, prevention of malaria in pregnancy and other infections; provision of holistic care to ensure normal progression of the baby and good health of the mother.

INTERVENTIONS:
Behavioral: gender-based violence screening, first-line support (LIVES) and reproductive coercion empowerment counseling (ARCHES) — Providers will (1) introduce routine client screening for GBV, including intimate partner violence, sexual violence, and reproductive coercion using a standardized screening form, in FP and ANC services,(2) for individuals disclosing GBV, provide first-line response-empathetic counseling, including listening, inquiring about experiences sensitively, and validating experiences, helping clients develop safety plans, and providing support; (3) regardless of disclosure of GBV, provide counseling and information, education and communication (IEC) materials on IPV, including reproductive coercion, and FP options, to both FP and ANC clients.
  Other Names: GBV screening, LIVES and ARCHES
  Arms: Treatment group

SUMMARY:
To pilot and evaluate the integration of first-line response to gender- based violence (GBV), particularly intimate partner violence (IPV), sexual violence and reproductive coercion, within family planning (FP) and antenatal care (ANC) services at public health facilities in Ebonyi and Sokoto states in Nigeria.

GBV first-line response in the health setting includes screening , empowerment counseling, safety planning, and support to connect to additional services needed.

DETAILED DESCRIPTION:
This study seeks to:

1. Assess effectiveness of an integrated service delivery model (integration of GBV first-line response and empowerment counseling in standard of care FP or ANC services) in reducing on-going experience of intimate partner violence (IPV) and increasing utilization of modern contraceptive methods among clients.

1a. Assess effectiveness of the intervention in reducing IPV, increasing utilization of modern contraceptive methods, and improving safety and self-efficacy among clients seeking interval FP services.

1b. Assess effectiveness of the intervention in reducing IPV and improving safety and self-efficacy to seek GBV care among clients seeking ANC services.

2. Explore factors influencing feasibility, acceptability and ability to implement GBV first-line response as part of FP and ANC services.

ELIGIBILITY:
Inclusion Criteria:

* Woman of reproductive age (18 to 49 years) seeking FP or ANC services at study sites
* Women who believe they are able to conceive (i.e. who have not undergone a tubal ligation, hysterectomy, or oophorectomy, or are menopausal) (for FP clients)
* Have a male partner they currently have sex with
* Have a mobile phone that can be safely used for re-contacting for follow-up surveys
* Do not have any accompanying male partners or family members aged 5 or above present

Exclusion Criteria:

* Any individuals that do not meet all of the above inclusion criteria or do not agree to participate in the study will be excluded from data collection.
* In addition, individuals with impaired cognitive abilities (I.e. unable to make decisions/respond to questions on their own without assistance by someone else)will also be excluded from the data collection.
* Finally, women who share a mobile phone with their partner/husband or another family member will also be excluded.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 1756 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in percentage of clients disclosing exposure to intimate partner or sexual violence in past 3 months | baseline to 3-months and 6-months post-intervention
  Disclosure will be defined by a positive response to either of the following questions:
  * Has your current partner ever slapped you, punched you, hit or kicked you, or done anything else to hurt you physically?
  * Has your current male partner ever forced you to have sex or do something sexual when you didn't want to?
Percentage of clients that report receiving a family planning method from healthcare provider | day of intervention

SECONDARY OUTCOMES:
Change in percentage of clients demonstrating family planning self efficacy, as measured by Contraceptive Self-Efficacy among women in sub-Saharan Africa (CSESSA) sub-scale | baseline to 3-months and 6-months post-intervention
  Family planning self-efficacy is a women's belief about her own ability to complete the actions necessary for successful family planning.
Change in demonstrated self-efficacy to access IPV services | baseline to 3-months and 6-months post-intervention
  Self-efficacy to access IPV services is an IPV survivor's confidence to develop and execute a plan when her partner becomes violent/ if her partner were to become violent. Self-efficacy will be defined by an affirmative response to the following questions:
  * I am confident that I could develop a plan for seeking help 'when my partner becomes violent/ if my partner were to become violent'
  * I am confident that I would be able to execute my plan 'in times when my partner becomes violent / if my partner were to become violent'.
Change in self-reported use of safety measures to protect respondent or her child/children from violence | baseline to 3-months and 6-months post-intervention
  Whether an IPV survivor has ever done any of the following to protect herself or her child/children for fear that her partner would become violent:
  * Identified a safe place to go in case she needs to leave her home ?
  * Identified a friend or relative to whom she could seek help?
  * Set aside some things she may need, such as clothes, documents in case she needs to leave in a hurry?
  * Set aside funds in case she needs to leave your home/partner?
  * Made a plan for what she would do with her child/children in case she needs to leave home?
Change in percentage of clients reporting experiences of reproductive coercion in 3 months prior to data collection | baseline to 3-months and 6-months post-intervention
  Reproductive coercion is behavior that interferes with the autonomous decision-making of a woman, with regards to reproductive health, including whether client felt pressured or forced by current partner to become pregnant or made it difficult to use family planning. Reproductive coercion will be defined by a positive response to either of the following questions:
  * Have you ever felt pressured or forced by your current partner to become pregnant when you did not want to be?
  * Has your current partner ever made it difficult for you to get family planning or to use family planning?

OTHER OUTCOMES:
Clients perception of quality of services provided | day of intervention
  Perception of service quality will be defined by a positive or negative response to the following question:
  • Has any provider from this clinic made you feel uncomfortable or treated you badly (e.g. insulted or disrespected you) for wanting to use or for using a family planning method?
Knowledge of intimate partner violence (IPV) and sexual violence (SV) related services | baseline to 3-months and 6-months post-intervention
  Knowledge will be defined as a positive response to whether client thinks a woman experiencing physical or sexual violence from her male partner could get help at specified services (health services, law enforcement, legal aid services, psychosocial support services, shelter/temporary accomodation, economic reintegration services).
Change in self-reported communication with partner about family planning | baseline to 3-months and 6-months post-intervention
  Couple communication about family planning will be defined by a positive response to the following question:
  • In the last 3 months, did you discuss whether to use a family planning method with your husbands/partner?
Change in self-reported communication with partner about birth plan | baseline to 3-months and 6-months post-intervention
  Couple communication about birth plan will be defined by a positive response to the following question:
  • In the past 3 months, did you discuss your birth plan with your partner?

CONTACTS AND LOCATIONS:
Overall Officials: Myra Betron, Principal Investigator — Jhpiego
Locations (40):
- Nigeria (40):
  - AZUIYIOKWU Health Center, Abakaliki, Ebonyi State
  - GMELINA Health Center, Abakaliki, Ebonyi State
  - NEW TIMBER SHADE Health Center, Abakaliki, Ebonyi State
  - AMAECHARA Primary Health Center, Afikpo North, Ebonyi State
  - Izeke Health Center, Afikpo North, Ebonyi State
  - NKAGBOGO NDEMIYI MDG Primary Health Center, Afikpo North, Ebonyi State
  - Owutu Primary Health Center, Afikpo South, Ebonyi State
  - Uwana Primary Health Center, Afikpo South, Ebonyi State
  - MDG Randa, Ebonyi, Ebonyi State
  - MCH Onueke, Ezza South, Ebonyi State
  - AZUNRAMURA Health Center, Ezza, Ebonyi State
  - Cottage Hospital, Ikwo, Ebonyi State
  - Echara Health Center, Ikwo, Ebonyi State
  - Item Health Center, Ikwo, Ebonyi State
  - Noyo Health Center, Ikwo, Ebonyi State
  - NDIOKOROUKWU Health Center, Ivo, Ebonyi State
  - Anike Health Center, Onicha, Ebonyi State
  - Okaria Health Center, Onicha, Ebonyi State
  - Oshiri Health Center, Onicha, Ebonyi State
  - GH Bodinga, Bodina, Sokoto State
  - Durbawa Primary Health Center, Dange Sguni, Sokoto State
  - Kwannawa Primary Health Center, Dange Sguni, Sokoto State
  - Ruga Dubu, Dange Sguni, Sokoto State
  - GH Gada, Gada, Sokoto State
  - Mamman Suka Primary Health Center, Gwadabawa, Sokoto State
  - Araba Health Center, Ilela, Sokoto State
  - Darna Sabon Gari Health Center, Ilela, Sokoto State
  - Garu, Ilela, Sokoto State
  - Gidan Chiwake Health Center, Ilela, Sokoto State
  - Gidan Hamma Health Center, Ilela, Sokoto State
  - Kalmalo, Ilela, Sokoto State
  - Rungumawar Gatti Health Center, Ilela, Sokoto State
  - Tozai Health Center, Ilela, Sokoto State
  - AKAEZEUKWU Health Center, Ivo, Sokoto State
  - Durbawa Primary Health Center, Kware, Sokoto State
  - Gan Gam Primary Health Center, Shagari, Sokoto State
  - Horo Primary Health Center, Shagari, Sokoto State
  - Kajiji Primary Health Center, Shagari, Sokoto State
  - Sanyinnawal Primary Health Center, Shagari, Sokoto State
  - Kaura Kimba Health Post, Wamako, Sokoto State

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uysal J, Carter N, Johns N, Boyce S, Liambila W, Undie CC, Muketo E, Adhiambo J, Gray K, Wendoh S, Silverman JG. Protocol for a matched-pair cluster control trial of ARCHES (Addressing Reproductive Coercion in Health Settings) among women and girls seeking contraceptive services from community-based clinics in Nairobi, Kenya. Reprod Health. 2020 May 27;17(1):77. doi: 10.1186/s12978-020-00916-9. PMID 32460786
- [Background] Pallitto C, Garcia-Moreno C, Stoeckl H, Hatcher A, MacPhail C, Mokoatle K, Woollett N. Testing a counselling intervention in antenatal care for women experiencing partner violence: a study protocol for a randomized controlled trial in Johannesburg, South Africa. BMC Health Serv Res. 2016 Nov 5;16(1):630. doi: 10.1186/s12913-016-1872-x. PMID 27814706
- [Background] Bacchu L, Mezey G, Bewley S. Women's perceptions and experiences of routine enquiry for domestic violence in a maternity service. BJOG. 2002 Jan;109(1):9-16. doi: 10.1111/j.1471-0528.2002.00514.x. PMID 11843378
- [Background] Boyle A, Jones PB. The acceptability of routine inquiry about domestic violence towards women: a survey in three healthcare settings. Br J Gen Pract. 2006 Apr;56(525):258-61. PMID 16611513
- [Background] McDonnell E, Holohan M, Reilly MO, Warde L, Collins C, Geary M. Acceptability of routine enquiry regarding domestic violence in the antenatal clinic. Ir Med J. 2006 Apr;99(4):123-4. PMID 16972587
- [Background] Waalen J, Goodwin MM, Spitz AM, Petersen R, Saltzman LE. Screening for intimate partner violence by health care providers. Barriers and interventions. Am J Prev Med. 2000 Nov;19(4):230-7. doi: 10.1016/s0749-3797(00)00229-4. PMID 11064226
- [Background] Hamberger L.K.; Guse C.; Boerger J.; Minsky D.; Pape D.; Folsom C. Evaluation of a Health Care Provider Training Program to Identify and Help Partner Violence Victims. Journal of Family Violence, Volume 19, Number 1, February 2004, pp. 1-11
- [Background] McNulty A, Andrews P, Bonner M. Can screening for domestic violence be introduced successfully in a sexual health clinic? Sex Health. 2006 Sep;3(3):179-82. doi: 10.1071/sh05056. PMID 17044223
- [Background] McNutt LA, Carlson BE, Rose IM, Robinson DA. Partner violence intervention in the busy primary care environment. Am J Prev Med. 2002 Feb;22(2):84-91. doi: 10.1016/s0749-3797(01)00407-x. PMID 11818176
- [Background] Taft A, Colombini M. Healthcare system responses to intimate partner violence in low and middle-income countries: evidence is growing and the challenges become clearer. BMC Med. 2017 Jul 12;15(1):127. doi: 10.1186/s12916-017-0886-5. PMID 28697810
- [Result] McFarlane JM, Groff JY, O'Brien JA, Watson K. Secondary prevention of intimate partner violence: a randomized controlled trial. Nurs Res. 2006 Jan-Feb;55(1):52-61. doi: 10.1097/00006199-200601000-00007. PMID 16439929
- [Result] Tiwari A, Leung WC, Leung TW, Humphreys J, Parker B, Ho PC. A randomised controlled trial of empowerment training for Chinese abused pregnant women in Hong Kong. BJOG. 2005 Sep;112(9):1249-56. doi: 10.1111/j.1471-0528.2005.00709.x. PMID 16101604
- [Result] Miller E, Decker MR, McCauley HL, Tancredi DJ, Levenson RR, Waldman J, Schoenwald P, Silverman JG. A family planning clinic partner violence intervention to reduce risk associated with reproductive coercion. Contraception. 2011 Mar;83(3):274-80. doi: 10.1016/j.contraception.2010.07.013. PMID 21310291
- [Result] Kiely M, El-Mohandes AAE, El-Khorazaty MN, Gantz MG. An integrated intervention to reduce intimate partner violence in pregnancy: a randomized controlled trial. Obstet Gynecol. 2010 Feb;115(2 Pt 1):273-283. doi: 10.1097/AOG.0b013e3181cbd482. PMID 20093899
- [Derived] Betron M, Bryce E, Obafemi S, Yusuf S, Abdullahi H, Ifemenam E, Dikeocha N, Maiakwai A, Kabir B, Oduenyi C. Effectiveness of a clinic-based counselling intervention on risk of experiencing intimate partner violence and reproductive coercion: a matched-pair cluster-controlled trial in Ebonyi and Sokoto, Nigeria. BMJ Glob Health. 2025 Oct 28;10(10):e016898. doi: 10.1136/bmjgh-2024-016898. PMID 41151831
- See also: World Health Organization. (2019). Caring for women subjected to violence: a WHO curriculum for training health-care providers. World Health Organization. — https://apps.who.int/iris/handle/10665/330084